CLINICAL TRIAL: NCT03337139
Title: Improving Weight Loss Maintenance by Using Digital Data Sharing to Provide Responsive Support and Accountability
Brief Title: FitLink: Improving Weight Loss Maintenance by Using Digital Data to Provide Support and Accountability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Office of Behavioral and Social Sciences Research (OBSSR) (NIH)
Responsible Party: Principal Investigator, Meghan Butryn, Principle Investigator, Drexel University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1611004954; R21DK112741 (NIH)
Record Dates: First submitted 2017-11-07; First posted 2017-11-08 (Actual); Results first posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Obesity; Overweight; Overweight and Obesity; Weight Loss
Keywords: Weight Loss; Obesity; Overweight; Behavioral Weight Loss
MeSH Terms: conditions — Obesity; Overweight; Weight Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle Modification (Active Comparator): Three months of standard, group-based behavioral treatment for weight loss and nine months of remote individual behavioral treatment based on self-report.
  Interventions: Behavioral: Gold Standard Behavior Therapy for Weight Loss; Behavioral: Standard Remote Behavior Therapy for Weight Loss
- Lifestyle Modification + Share (Experimental): Three months of standard, group-based behavioral treatment for weight loss and nine months of remote individual behavioral treatment based on digital data shared with clinicians.
  Interventions: Behavioral: Gold Standard Behavior Therapy for Weight Loss; Behavioral: Digital Data Sharing Behavior Therapy for Weight Loss

INTERVENTIONS:
Behavioral: Gold Standard Behavior Therapy for Weight Loss — Group-based behavioral treatment for weight loss, with a standard emphasis on diet (65% of session) and physical activity goals (25% of session). Other weight loss behaviors such as self monitoring will be covered in the remaining time (10% of session). Participants will be asked to utilize digital monitoring devices for physical activity, weight, and diet. Coaches will not have access to the digital data that participants provide on physical activity, weight, and diet monitoring devices.
Behavioral: Standard Remote Behavior Therapy for Weight Loss — Individual, monthly, brief phone calls with coach and weekly text messages. The content of these calls and messages will be determined by participant self-report. Coaches will not have access to the digital data that participants provide on physical activity, weight, and diet monitoring devices.
  Arms: Lifestyle Modification
Behavioral: Digital Data Sharing Behavior Therapy for Weight Loss — Individual, monthly, brief phone calls with coach and weekly text messages. The content of these calls and messages will be determined by the digital data that has been shared with the coach from physical activity, weight, and diet monitoring devices.
  Arms: Lifestyle Modification + Share

SUMMARY:
Most adults in the U.S. are overweight or obese and find maintenance of weight loss difficult. This study is designed to aid in the development of a lifestyle modification program that can facilitate weight loss maintenance, without requiring long-term visits to a clinic for maintenance treatment.

DETAILED DESCRIPTION:
In a lifestyle modification program, contact with an interventionist (e.g., weight loss coach) creates a sense of supportive accountability that can facilitate behavior change and weight loss. Sustaining a strong sense of supportive accountability after face-to-face intervention contact ends has the potential to improve outcomes during the notoriously difficult weight loss maintenance period. One innovative way of facilitating supportive accountability is providing participants with digital tools that objectively measure weight and physical activity and track food intake in real-time, making the data from those tools automatically and continuously available to coaches, and designing the timing and content of intervention contacts such that they are responsive to the shared data. Although tools that allow for data sharing from sensors and Internet-based applications are readily available, the ways in which they are integrated into intervention contacts in a lifestyle modification program are not yet optimized, and research has not systematically evaluated the effect of data sharing on behavior. Overweight and obese participants (n = 90) will be recruited from the community for a small randomized controlled trial in order to test the feasibility, acceptability, efficacy, and mechanisms of action of a lifestyle modification intervention enhanced with data sharing. In weeks 1-12 of the program (i.e., Phase I), all participants will attend 12 weekly, face-to-face, group-based behavioral treatment sessions to induce weight loss. Participants will be provided with a wireless body weight scale, physical activity sensor, and digital food record app and instructed to use them daily use for self-monitoring purposes. In Phase II (weeks 13-52), participants will be randomly assigned to the standard (LM) or enhanced version of remote lifestyle modification (LM+SHARE). Neither condition will have face-to-face intervention contact during Phase II; remote intervention contact will consist of brief phone calls and text messages provided by the participant's coach. Participants in both conditions will be prescribed continued daily use of the three self-monitoring devices. In the standard LM condition, no digital data from these devices will be directly shared with coaches; intervention encounters will be informed only by the infrequent, delayed self-report of participants (which is the current standard of long-term obesity care), and timing of text messages will be fixed. In LM+SHARE, the digital tools will automatically and continuously transmit body weight, physical activity, and food record data to the coach. In LM+SHARE, supportive accountability will be enhanced in three ways: 1) participants will receive automated alerts after coaches view their data, 2) timing of personalized text messages from coaches will be responsive to clinically notable change in weight, physical activity, calorie intake, or use of scale, physical activity sensor, or food record tool, and 3) content of the text messages and phone calls will be informed by the digital data the coach has viewed, as well as the expectation that the coach will continue viewing data in order to provide ongoing support. Assessments will be completed at 0, 12, 26, and 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-70 years with a BMI of 25-45 kg/m2 and weight <160 kg
* Access to a smartphone
* Satisfactory completion of all enrollment procedures
* Ability to engage in physical activity (i.e. can walk at least 2 blocks without stopping for rest)

Exclusion Criteria:

* Medical condition (i.e. acute coronary syndrome, type 1 diabetes, renal failure) or psychiatric condition (i.e. active substance abuse, eating disorder) that may:

  * Pose a risk to the participant during the intervention
  * Cause a change in weight
  * Limit ability to comply with the behavioral recommendations of the program
* Pregnant or planning pregnancy in the next 1 year
* Planned move out of the Philadelphia area during the data collection period
* Use of a pacemaker (incompatible with wireless scale technology)
* Recently began or changed the dosage of a medication that can cause significant change in weight
* History of bariatric surgery
* Weight loss of > 10% in the previous 3 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meghan L Butryn, Ph.D., Principal Investigator — Drexel University
Locations (1):
- Drexel University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Butryn ML, Martinelli MK, Crane NT, Godfrey K, Roberts SR, Zhang F, Forman EM. Counselor Surveillance of Digital Self-Monitoring Data: A Pilot Randomized Controlled Trial. Obesity (Silver Spring). 2020 Dec;28(12):2339-2346. doi: 10.1002/oby.23015. Epub 2020 Oct 23. PMID 33098278
- [Derived] Schumacher LM, Martinelli MK, Convertino AD, Forman EM, Butryn ML. Weight-Related Information Avoidance Prospectively Predicts Poorer Self-Monitoring and Engagement in a Behavioral Weight Loss Intervention. Ann Behav Med. 2021 Mar 16;55(2):103-111. doi: 10.1093/abm/kaaa034. PMID 32491152

RESULTS

PARTICIPANT FLOW:
Period: Phase I
Arm/Group | Lifestyle Modification | Lifestyle Modification + Share
Started | 87 | 0 (There were not two conditions in Phase I: all participants received standard group LM treatment.)
Completed | 77 | 0
Not Completed | 10 | 0
Not completed — Withdrawal by Subject | 10 | 0
Period: Phase II
Arm/Group | Lifestyle Modification | Lifestyle Modification + Share
Started | 38 | 39
26 Week Assessment | 34 | 37
Completed | 33 | 36
Not Completed | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lifestyle Modification | Lifestyle Modification + Share | Total
Number analyzed (Participants) | 38 | 39 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.71 (13.33) | 49.84 (13.56) | 50.77 (13.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 32 | 62
  Male | 8 | 7 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 36 | 38 | 74
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 15 | 28
  White | 19 | 22 | 41
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 38 | 39 | 77

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight
Description: Objectively measured in the research clinic at each time point on a scale. Reported as weight change in kg, where negative numbers reflect weight loss and positive numbers reflect weight gain.
Time Frame: 0, 13, 26, 52 weeks
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Lifestyle Modification | Lifestyle Modification + Share
Number analyzed (Participants) | 38 | 39
kg
  13 weeks | -5.78 (4.79) | -5.80 (4.01)
  26 weeks | -1.76 (2.81) | -1.54 (2.83)
  52 weeks | 1.98 (3.22) | 0.06 (4.16)
Statistical Analysis 1: Comparison: Lifestyle Modification vs Lifestyle Modification + Share; Comparing groups on 13 week weight loss, prior to randomization; Test type: Superiority; p = .98, ANCOVA — A priori threshold for statistical significance was p <.05
Statistical Analysis 2: Comparison: Lifestyle Modification vs Lifestyle Modification + Share; Comparing groups on 26 week weight loss; Test type: Superiority; p = .75, ANCOVA — A priori threshold for statistical significance was p <.05; Controlling for Phase I weight loss
Statistical Analysis 3: Comparison: Lifestyle Modification vs Lifestyle Modification + Share; Comparing groups on 52 week weight loss; Test type: Superiority; p = .02, ANCOVA — A priori threshold for statistical significance was p<.05; Controlling for Phase I weight loss

2. Primary Outcome: Change in Physical Activity
Description: Objectively measured using wGT3X-BT accelerometers from Actigraph. Minutes/week of moderate-to-vigorous physical activity (MVPA).
Time Frame: 13, 52 weeks
Measure: Mean (Standard Deviation); unit: min per week of bouted MVPA
Arm/Group | Lifestyle Modification | Lifestyle Modification + Share
Number analyzed (Participants) | 38 | 39
min per week of bouted MVPA
  13 weeks | 173.62 (137.16) | 125.86 (134.16)
  52 weeks | 94.15 (99.39) | 101.68 (98.16)
Statistical Analysis 1: Comparison: Lifestyle Modification vs Lifestyle Modification + Share; Comparing groups on 13 week MVPA; Test type: Superiority; p = .12, ANCOVA — A priori threshold for statistical significance was p <.05
Statistical Analysis 2: Comparison: Lifestyle Modification vs Lifestyle Modification + Share; Comparing groups on 52 week MVPA; Test type: Superiority; p = .16, ANCOVA — A priori threshold for statistical significance was p<.05; Controlling for changes in Phase I MVPA

3. Primary Outcome: Number of Participants Retained
Description: Feasibility and acceptability metric of retention.
Time Frame: 26, 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Lifestyle Modification | Lifestyle Modification + Share
Number analyzed (Participants) | 38 | 39
Participants
  26 weeks | 34 | 37
  52 weeks | 33 | 36
Statistical Analysis 1: Comparison: Lifestyle Modification vs Lifestyle Modification + Share; Comparing groups on 26 week retention rates; Test type: Superiority; p = .43, Fisher Exact — A priori threshold for statistical significant was p<.05
Statistical Analysis 2: Comparison: Lifestyle Modification vs Lifestyle Modification + Share; Comparing groups on 52 week retention rates; Test type: Superiority; p = .48, Fisher Exact — A priori threshold for statistical significance was p<.05

4. Primary Outcome: Number of Completed Treatment Contacts
Description: Feasibility and acceptability metric of completed treatment contacts (phone calls and text messages).
Time Frame: 52 weeks
Measure: Mean (Standard Deviation); unit: number completed
Arm/Group | Lifestyle Modification | Lifestyle Modification + Share
Number analyzed (Participants) | 38 | 39
number completed
  Phone Calls | 7.37 (1.55) | 7.20 (1.79)
  Text Messages | 30.50 (3.85) | 29.67 (5.94)
Statistical Analysis 1: Comparison: Lifestyle Modification vs Lifestyle Modification + Share; Comparing groups on phone calls completed in Phase II (52 weeks); Test type: Superiority; p = .64, Permutation test — A priori threshold of statistical significance was p<.05; Permutation test (nonparametric test) was chosen due to the violation of t-test assumptions in the data set
Statistical Analysis 2: Comparison: Lifestyle Modification vs Lifestyle Modification + Share; Comparing groups on text messages completed in Phase II (52 weeks); Test type: Superiority; p = .499, Permutation test — A priori threshold for statistical significance was p<.05; Permutation test (nonparametric test) was chosen due to the violation of t-test assumptions in the data set

5. Primary Outcome: Treatment Acceptability Questionnaire (TAQ)
Description: Feasibility and acceptability metric of scores on the TAQ. Items on the TAQ consisted of 11 questions on a 7 point Likert scale asking about helpfulness and acceptability of treatment components. Items are summed to yield a total score that can range from 11-77 with higher numbers indicated higher acceptability.
Time Frame: 52 weeks
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Lifestyle Modification | Lifestyle Modification + Share
Number analyzed (Participants) | 38 | 39
score | 65.62 (8.43) | 65.95 (7.76)
Statistical Analysis 1: Comparison: Lifestyle Modification vs Lifestyle Modification + Share; Comparing groups on TAQ scores at 52 weeks; Test type: Superiority; p = .86, Permutation test — A priori threshold for statistical significance was p<.05; Permutation test (nonparametric test) was chosen due to the violation of t-test assumptions in the data set

6. Secondary Outcome: Self-monitoring Engagement
Description: Use of digital devices; percent of days during which weight, food, and steps were counted in Phase II. Percent calculated for each group (LM vs. LM+Share) and not for individual participants. We determined percent to be the metric that would be most easily interpreted and it accounted for any possible variability in total number of days of observations.
Time Frame: 13-52 weeks
Measure: Number; unit: percent days self-monitoring occurred
Arm/Group | Lifestyle Modification | Lifestyle Modification + Share
Number analyzed (Participants) | 38 | 39
percent days self-monitoring occurred
  Weight | 43 | 58
  Eating | 41 | 67
  Physical Activity | 79 | 80
Statistical Analysis 1: Comparison: Lifestyle Modification vs Lifestyle Modification + Share; Comparing groups on percent days of self-monitoring of weight during Phase II; Test type: Superiority; p = .002, ANCOVA — A priori threshold for statistical significance was p<.05; Controlling for Phase I engagement in self-monitoring
Statistical Analysis 2: Comparison: Lifestyle Modification vs Lifestyle Modification + Share; Comparing groups on percent days of self-monitoring of eating during Phase II; Test type: Superiority; p = .001, ANCOVA — A priori threshold for statistical significance was p<.05; Controlling for Phase I engagement in self-monitoring
Statistical Analysis 3: Comparison: Lifestyle Modification vs Lifestyle Modification + Share; Comparing groups on percent days of self-monitoring of physical activity during Phase II; Test type: Superiority; p = .25, ANCOVA — A priori threshold for statistical significance was p<.05; Controlling for Phase I engagement in self-monitoring

7. Secondary Outcome: Perceived Accountability
Description: Change in "Perceptions of Accountability" subscale of the Supportive Accountability Scale. The measure used was a 10-item scale on which participants rated the extent to which they agreed with statements on a 7-point likert scale. A total score was generated by summing scores from individual items. Total scores ranged from 10-70 with higher scorings indicating higher perceived accountability. The outcome measure reported here is the change in total score on this measure (decrease) across Phase II where a negative score reflects a decrease in perceived accountability.
Time Frame: 52 weeks
Measure: Mean (Standard Deviation); unit: unit change
Arm/Group | Lifestyle Modification | Lifestyle Modification + Share
Number analyzed (Participants) | 38 | 39
unit change | 8.28 (15.25) | 6.88 (16.05)
Statistical Analysis 1: Comparison: Lifestyle Modification vs Lifestyle Modification + Share; Comparing groups on changes in perceived accountability during Phase II; Test type: Superiority; p = .005, ANCOVA — A priori threshold for statistical significance was p<.05; Controlling for Phase I perceived supportive accountability

ADVERSE EVENTS:
Time Frame: 52 weeks (entire study period)
Arm/Group | Lifestyle Modification | Lifestyle Modification + Share
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/39
Other Adverse Events (participants affected / at risk) | 0/38 | 3/39
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lifestyle Modification (N=38) | Lifestyle Modification + Share (N=39)
Gallstones (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lightheadedness (Vascular disorders) | 0 (0) | 1 (1) — Due to blood pressure medication
Kidney Stone (Renal and urinary disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Low proportion of men and adults over age 70 limits generalizability; calls and texts were not qualitatively analyzed nor rated for treatment fidelity; length of each telephone session was not measured; it is unknown to what extent participants shared device data with friends/family/other participants and threatened contamination; low power.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-30): https://cdn.clinicaltrials.gov/large-docs/39/NCT03337139/Prot_SAP_000.pdf